CLINICAL TRIAL: NCT04543812
Title: A Phase 3 Study of PBF-1681 Comprising a 16-week, Placebo-controlled, Double-blind Randomized Period and an 8-week, Open-label Extension Period for the Treatment of Iron Deficiency Anemia in Patients With Non-Dialysis Dependent CKD
Brief Title: PBF-1681 (Ferric Citrate) for the Treatment of IDA in Patients With NDD-CKD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Panion & BF Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PBB00601
Record Dates: First submitted 2020-09-02; First posted 2020-09-10 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Anemia of Chronic Kidney Disease
Keywords: Ferric Citrate; Anemia; Chronic Kidney Disease
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — ferric citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PBF-1681 (ferric citrate) (Experimental): PBF-1681 (ferric citrate) will be dosed two times a day with the 2 largest meals (preferred) or three times a day with meals.
  Interventions: Drug: Ferric citrate
- Placebo (Placebo Comparator): Matching placebo will be dosed two times a day with the 2 largest meals (preferred) or three times a day with meals.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ferric citrate — Ferric citrate will be provided as a 1g tablet. All intervention doses will be based on hemoglobin levels.
  Arms: PBF-1681 (ferric citrate)
Drug: Placebo — Matching placebo will be provided as a 1g tablet. All intervention doses will be based on hemoglobin levels.
  Arms: Placebo

SUMMARY:
To assess the safety and effectiveness of PBF-1681 for the treatment of Iron Deficiency Anemia in patients with Non-Dialysis Dependent Chronic Kidney Disease.

DETAILED DESCRIPTION:
This is a Phase 3, 24-week, multicenter study in Taiwan, comprising a 16-week, randomized, double-blind, placebo-controlled period ("Randomized Period"), followed by an 8-week open-label extension period, where all subjects receive PBF-1681 (ferric citrate) ("Extension Period"). The study will consist of 10 visits over a period of 24 weeks. There will be a screening period of up to 14 days. Approximately 200 subjects will be randomized into the Randomized Period in a 1:1 ratio to receive either PBF-1681 or matching placebo, at baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women ≥18 years of age at screening.
2. CKD with eGFR <60 mL/min at screening using the 4-variable Modification of Diet in Renal Disease equation, where up to 20% of subjects with eGFR <15 mL/min are allowed.
3. Hgb ≥9.0 g/dL and ≤11.5 g/dL at screening.
4. Serum ferritin <300 ng/mL and TSAT <30% at screening.
5. Serum iPTH ≤600 pg/mL at screening.
6. Must consume minimally 2 meals per day.
7. Willing to give written informed consent.
8. Women may be enrolled if they are:

   1. Documented to be surgically sterile or postmenopausal (amenorrhea >1 year and follicle-stimulating hormone ≥30 mU/mL), or
   2. Practicing true abstinence for at least 28 days prior to study drug administration until 30 days after study drug administration and having a negative serum pregnancy test at screening, or
   3. Using 2 forms of highly effective contraception, out of which 1 should be a physical barrier (condom or diaphragm), and another method such as adequate hormonal method (eg, contraceptive implants, injectables, oral contraceptives) or non-hormonal methods (eg, intrauterine device, spermicidals) from screening or at least 2 weeks prior to study drug administration (whichever is earlier) until 30 days after the study drug administration and having a negative serum pregnancy test at screening.

Exclusion Criteria:

1. Cause of anemia other than iron deficiency.
2. Serum phosphate <3.0 mg/dL at screening.
3. IV iron administered within 4 weeks of the start of screening.
4. ESA administered within 4 weeks of the start of screening.
5. Blood transfusion within 4 weeks of the start of screening.
6. Liver enzymes (alanine aminotransferase [ALT]/aspartate aminotransferase [AST]) >3 times upper limit of normal (ULN) at screening.
7. Symptomatic GI bleeding or symptomatic inflammatory bowel disease within 12 weeks of the start of screening.
8. Concurrent GI diseases assessed by Investigators to be inappropriate for the study, eg, acute peptic ulcer, chronic ulcerative colitis, and regional enteritis.
9. Active infection requiring systemic antimicrobial treatment such as antibiotics, antiviral, or antifungals at screening.
10. Concomitant or prior malignancy, except non-melanoma skin cancer or disease-free for ≥2 years after curative therapy.
11. Subjects with known allergic reaction to previous oral iron therapy.
12. Subjects who were intolerant to oral iron therapy.
13. History of hemochromatosis.
14. Scheduled kidney transplant or initiation of dialysis planned within 24 weeks of the start of screening.
15. Planned surgery or hospitalization (anticipated to last >72 hours) during the Randomized Period of the study other than dialysis access-related surgery.
16. Any other medical condition that, in the Investigators' opinion, may disturb subject's completion or optimal participation of the study, act as a significant confounding variable, or carry significant risks to a subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Hemoglobin (Hgb) | 16 weeks
  The mean change from baseline to the end of the Randomized Period in Hgb.

SECONDARY OUTCOMES:
Proportion of Subjects with ≥1.0 g/dL Hgb Increase at any time point | 16 weeks
  The proportion of subjects achieving an increase in Hgb of ≥1.0 g/dL at any time point between baseline and the end of the 16-week Randomized Period.
Transferring saturation (TSAT) | 16 weeks
  The mean change from baseline to the end of the Randomized Period in TSAT.
Ferritin | 16 weeks
  The mean change from baseline to the end of the Randomized Period in ferritin.
Serum Phosphate | 16 weeks
  The mean change from baseline to the end of the Randomized Period in serum phosphate.
Sustained increase in Hgb of ≥0.75 g/dL | 16 weeks
  The proportion of subjects achieving a sustained increase in Hgb of ≥0.75 g/dL from baseline over any 4-week interval during the Randomization Period.

OTHER OUTCOMES:
Serum calcium | 16 weeks
  The mean change from baseline to the end of the Randomized Period in serum calcium.
Serum bicarbonate | 16 weeks
  The mean change from baseline to the end of the Randomized Period in serum bicarbonate.
Serum iron | 16 weeks
  The mean change from baseline to the end of the Randomized Period in serum iron.
Unsaturated iron binding capacity (UIBC) | 16 weeks
  The mean change from baseline to the end of the Randomized Period in UIBC.
Total iron binding capacity (TIBC) | 16 weeks
  The mean change from baseline to the end of the Randomized Period in TIBC.
Hematocrit | 16 weeks
  The mean change from baseline to the end of the Randomized Period in hematocrit.
Intact parathyroid hormone (iPTH) | 16 weeks
  The mean change from baseline to the end of the Randomized Period in iPTH.
Fibroblast growth factor 23 (intact and C-terminal) | 16 weeks
  The mean change from baseline to the end of the Randomized Period in FGF23 (intact and C-terminal).
Serum aluminum | 16 weeks
  The mean change from baseline to the end of the Randomized Period in serum aluminum.
Sustained increase in Hgb | 16 weeks
  The proportion of subjects achieving a sustained increase in Hgb of ≥0.75 g/dL from baseline over any 4-week interval during the Randomized Period, provided that an increase in Hgb of ≥1.0 g/dL had occurred during that 4-week interval
Increase in Hgb of ≥1.0 g/dL | 16 weeks
  Time (in days) to first increase in Hgb of ≥1.0 g/dL from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Mei-I Wu, MD, PhD, Study Chair — Department of Internal Medicine, Taipei Medical University-Shuang Ho Hospital
Locations (12):
- Taiwan (12):
  - Division of Nephrology, Department of Internal Medicine, Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Division of Nephrology, Department of Internal Medicine, Kaohsiung Chang-Gung Memorial Hospital, Kaohsiung City
  - Division of Nephrology, Department of Internal Medicine, Keelung Chang Gung Memorial Hospital, Keelung
  - Division of Nephrology, Department of Internal Medicine, Far East Memorial Hospital, New Taipei City
  - Division of Nephrology, Department of Internal Medicine, China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Department of Integrated Diagnostics and Therapeutics, National Taiwan University Hospital, Taipei
  - Division of Nephrology, Department of Internal Medicine, Taipei Veterans General Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Municipal Wanfang Hospital, Taipei
  - Division of Nephrology, Department of Internal Medicine, Taipei Medical University-Shuang Ho Hospital, Taipei County
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District

IPD SHARING:
Plan to Share IPD: No